CLINICAL TRIAL: NCT05780125
Title: Effectiveness of Different Fibrinogen Preparations in Restoring Clot Firmness
Acronym: EDIPORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director of the Cardiovascular Anesthesia and Intensive Care Department, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EDIPORE
Record Dates: First submitted 2023-02-22; First posted 2023-03-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hypofibrinogenemia; Surgical Blood Loss; Bleeding; Cardiac Disease; Surgery
Keywords: hypofibrinogenemia; cardiac surgery; postoperative bleeding
MeSH Terms: conditions — Afibrinogenemia; Blood Loss, Surgical; Hemorrhage; Heart Diseases; Postoperative Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computerized system generated a randomization sequence, and then sealed envelopes containing the drug assigned was prepared. The randomization ratio of the treatment arms was 1:1. An unblinded biologist (E.B.) was in charge of running the ROTEM® tests, randomization, drug preparation, and masking, and its delivery to the operating room. The attending anesthesiologist, the surgical staff, and the medical staff in the ICU and ward were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FibCLOT (Experimental): Patients randomized to the FibCLOT arm will receive 30 mg/kg, approximated to the closest between 2 and 3 grams, of FibCLOT (LFB, Puteaux, France).
  Interventions: Drug: FibCLOT
- RiaSTAP (Active Comparator): Patients randomized to the RiaSTAP arm will receive 30 mg/kg, approximated to the closest between 2 and 3 grams, of RiaSTAP (King of Prussia, PA, USA).
  Interventions: Drug: RiaSTAP

INTERVENTIONS:
Drug: FibCLOT — 30 mg/kg of FibCLOT (rounded up to the nearest 2 or 3 grams) after protamine administration
  Other Names: Human Fibrinogen concentrate
  Arms: FibCLOT
Drug: RiaSTAP — 30 mg/kg of RiaSTAP (rounded up to the nearest 2 or 3 grams) after protamine administration
  Other Names: Human Fibrinogen concentrate
  Arms: RiaSTAP

SUMMARY:
Fibrinogen concentrate is produced by different manufacturers using different purification technologies. The products available in Italy are three: RiaSTAP (CSL Behring), FIBRYGA (Octapharma), and FibCLOT (LFB). RiaSTAP and FIBRYGA are sold in 1-gram vials, and FibCLOT - in 1.5-gram vials. A recent in vitro study assessed how these products affected the clot firmness measured by the ROTEM FIBTEM maximum clot firmness (MCF) parameter. In vitro conditions, FibCLOT was verified to be the most efficient in increasing clot firmness.

The present study is aimed to assess, in a series of patients undergoing cardiac surgery with cardiopulmonary bypass, the hypothesis that the FibCLOT fibrinogen is superior to the RiaSTAP fibrinogen in increasing the FIBTEM MCF parameter in a clinical model of bleeding (postoperative bleeding after complex cardiac surgery).

DETAILED DESCRIPTION:
The Effectiveness of DIfferent fibrinogen PreparatiOns in Restoring clot firmness (EDIPO RE) is a pragmatic, double-blinded, randomized controlled trial testing the hypothesis that FibCLOT is superior to RiaSTAP in restoring fibrinogen-dependent clot firmness in cardiac surgery acquired hypofibrinogenemia.

A randomization sequence was generated by a computerized system, and then sealed envelopes containing the drug assigned were prepared. The randomization ratio of the treatment arms was 1:1. An unblinded biologist was in charge of running the ROTEM® tests, randomization, drug preparation, and masking, and its delivery to the operating room. The attending anesthesiologist, the surgical staff, and the medical staff in the ICU and ward were blinded.

After protamine administration, if microvascular bleeding was observed or suspected, POC testing, including ROTEM® EXTEM and FIBTEM, was run. If FIBTEM MCF was lower than 10 mm, the patient was randomly allocated to receive a dose of RiaSTAP® or FibCLOT® of 30 mg/kg, approximated to the closest between 2 or 3 grams. If no sign of ongoing bleeding was present, or FIBTEM MCF was 10 mm or higher the patient was considered screen failure and excluded from further observation.

Forty patients were randomized to receive the assigned treatment.

Fibrinogen was administrated intravenously by infusion at a rate of approximately 20 ml/min. Ten minutes after fibrinogen administration a second test was performed with ROTEM® EXTEM and FIBTEM tests to record the change of the parameters due to fibrinogen supplementation. No other hemostatic drugs nor transfusions, outside the study drug, were administered between the first and the second testing. In case of ongoing intra- or postoperative bleeding, after the second testing, all the hemostatic corrections were allowed and guaranteed by our institutional protocol for postoperative bleeding management, which includes the following step-by-step interventions:

* 30-50 mg of additional protamine for the correction of residual heparin, if the CT at INTEM exceeded 20% of the CT at HEPTEM;
* Additional fibrinogen concentrate, if FIBTEM MCF < 10 mm or Clauss fibrinogen < 150 mg dL-1;
* Platelet concentrates if P2Y12 receptor inhibitors were discontinued not later than 7 days, a postoperative ADP test at Multiplate® aggregometry < 12 U, or a postoperative platelet count measured or presumed from preoperative count <100,000 cells/µL;
* 4-factors prothrombin complex concentrate (PCC, Pronativ, Octapharma, Lachen, Switzerland) 20 IU kg-1 if EXTEM CT > 100 s (after correction of fibrinogen and platelet values) or INR > 1,5.

Preoperative, and perioperative data and details of postoperative outcomes were retrieved from our institutional database and patients' medical charts, including demographics, preoperative risk factors, procedure details, postoperative bleeding and transfusions, intensive care unit (ICU), and hospital stay duration. For the study, the following additional data have been collected: preoperative fibrinogen, platelet count, coagulation parameters (prothrombin time, PT; international normalized ratio, INR; activated partial thromboplastin time, aPTT), post protamine EXTEM CT and MCF and FIBTEM MCF; post-fibrinogen supplementation EXTEM CT and MCF and FIBTEM MCF; fibrinogen, platelet count and coagulation at the ICU arrival.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery with cardiopulmonary bypass;
* complex cardiac surgery (coronary artery bypass graft + valve repair/replacement; double/triple valve repair/replacement; ascendant aorta surgery);
* written consent to participate;

Exclusion Criteria:

* urgent or emergent cardiac surgery;
* known hypersensitivity to the active principle or to one of the excipients of the study drugs;
* coagulation disorders, known or presumable from anamnesis;
* known hepatopathy;
* known risk of thrombosis or disseminated intravascular coagulation;
* participation in another clinical study where an experimental product has been administered within 30 days from the day of the inclusion in the study;
* whatever clinical condition that, in the opinion of the investigator, makes the patients not suitable to the experimentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
FIBTEM MCF (mm) | Within 10 minutes after protamine administration
  Fibrinogen contribution to the clot firmness measured by ROTEM device, as maximum clot firmness parameter).
FIBTEM CT and CFT (sec) | Within 10 minutes after protamine administration
  Fibrinogen contribution to the clot firmness measured by ROTEM device, as time required for clot formation (CT, clotting time, and CFT, clot formation time).
EXTEM CT and CFT (sec) | Within 10 minutes after protamine administration
  Time required for the overall clot formation on the extrinsic pathway of coagulation ( CT, clotting time, and CFT, clot formation time).

SECONDARY OUTCOMES:
Postoperative bleeding | 12 and 24 hours after surgery
  Amount of postoperative bleeding measured by the cardiac drainages
Incidence of moderate/severe bleeding | 12 hours after surgery
  Number of cases of moderate or severe bleeding, as defined by the Universal Definition of Perioperative bleeding
Incidence of transfusion | 12 and 24 hours after surgery
  Number of cases requiring the transfusion of red blood cells and platelet concentrates

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranucci M, Baryshnikova E. Fibrinogen supplementation after cardiac surgery: insights from the Zero-Plasma trial (ZEPLAST). Br J Anaesth. 2016 May;116(5):618-23. doi: 10.1093/bja/aev539. Epub 2016 Feb 17. PMID 26893405
- [Background] Stolt H, Shams Hakimi C, Singh S, Jeppsson A, Karlsson M. A comparison of the in vitro effects of three fibrinogen concentrates on clot strength in blood samples from cardiac surgery patients. Acta Anaesthesiol Scand. 2021 Nov;65(10):1439-1446. doi: 10.1111/aas.13967. Epub 2021 Sep 1. PMID 34368944
- [Background] Scolletta S, Simioni P, Campagnolo V, Celiento M, Fontanari P, Guadagnucci A, Guarracino F, Haxhiademi D, Paniccia R, Simeone F, Ranucci M; Granducato Research Group. Patient blood management in cardiac surgery: The "Granducato algorithm". Int J Cardiol. 2019 Aug 15;289:37-42. doi: 10.1016/j.ijcard.2019.01.025. Epub 2019 Jan 11. PMID 30711263
- [Background] Tibi P, McClure RS, Huang J, Baker RA, Fitzgerald D, Mazer CD, Stone M, Chu D, Stammers AH, Dickinson T, Shore-Lesserson L, Ferraris V, Firestone S, Kissoon K, Moffatt-Bruce S. STS/SCA/AmSECT/SABM Update to the Clinical Practice Guidelines on Patient Blood Management. J Cardiothorac Vasc Anesth. 2021 Sep;35(9):2569-2591. doi: 10.1053/j.jvca.2021.03.011. Epub 2021 Jun 30. No abstract available. PMID 34217578
- [Background] Dyke C, Aronson S, Dietrich W, Hofmann A, Karkouti K, Levi M, Murphy GJ, Sellke FW, Shore-Lesserson L, von Heymann C, Ranucci M. Universal definition of perioperative bleeding in adult cardiac surgery. J Thorac Cardiovasc Surg. 2014 May;147(5):1458-1463.e1. doi: 10.1016/j.jtcvs.2013.10.070. Epub 2013 Dec 9. PMID 24332097
- [Derived] Baryshnikova E, Aloisio T, Di Dedda U, Anguissola M, Barbaria A, Caravella G, Ranucci M. A Randomized Controlled Trial Comparing Effectiveness of Different Fibrinogen Preparations in Restoring Clot Firmness. Anesth Analg. 2025 Apr 1;140(4):966-973. doi: 10.1213/ANE.0000000000007201. Epub 2024 Oct 9. PMID 39383100